CLINICAL TRIAL: NCT05151848
Title: An Open-label，Randomized, Controlled, Multicenter Study of Adalimumab and Tofacitinib in the Treatment of Active Takayasu Arteritis
Brief Title: Comparison of Adalimumab and Tofacitinib in the Treatment of Active Takayasu Arteritis
Acronym: ADATOFTAK
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese SLE Treatment And Research Group (Other)
Responsible Party: Principal Investigator, Xinping Tian, Professor of Medicine, Chinese SLE Treatment And Research Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSTAR-007
Record Dates: First submitted 2021-11-06; First posted 2021-12-09 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Takayasu Arteritis
MeSH Terms: conditions — Takayasu Arteritis | interventions — Adalimumab; tofacitinib

STUDY DESIGN:
Intervention Model Description: open-label, multicenter,randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adalimumab group (Experimental): Adalimumab 40mg injected subcutaneously every 2 weeks for 78 weeks.
  Interventions: Drug: Adalimumab Injection
- Tofacitinib 5MG group (Active Comparator): Tofacitinib 5mg BID taken orally for 78 weeks.
  Interventions: Drug: Tofacitinib 5 MG

INTERVENTIONS:
Drug: Adalimumab Injection — Adalimumab Injection injected subcutaneously every other week for 78 weeks
  Other Names: An-jian-ning
  Arms: Adalimumab group
Drug: Tofacitinib 5 MG — Tofacitinib 5 MG BID taken orally for 78 weeks
  Other Names: An-shu-zheng
  Arms: Tofacitinib 5MG group

SUMMARY:
This is a prospective,open-labelled,multi-center,randomized clinical trial.It compares the clinical efficacy and safety of there 2 drugs in the treatment of relapse active Takayasu's arteritis patients.

DETAILED DESCRIPTION:
In this study, 100 relapse Takayasu's arteritis patients will be enrolled. Patients are randomized into the adalimumab treatment group and tofacitinib treatment.Patients will also be treated with reduced dose of glucocorticoid at the same time. The primary end point is the percentage of patients who are in complete response at week 12 and maintain in complete response at week 78.

The efficacy will be evaluated at week 12, 24, 36, 52 and 78. If the patient does not respond to one drug at week 24, then the investigator will shift the treatment to another intervention. Safety is also monitored during the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged between 18-65 years old;
2. Fulfilled the classification criteria of Takayasu's arteritis by ACR 1990;
3. relapse active TAK: defined by the definition of active disease in the recommendations released by EULAR in 2018;
4. Patients who signed the informed consent form.

Exclusion Criteria:

1. Patients who failed or intolerant to either adalimumab or tofacitinib;
2. patients with severe liver disease defined by the serum ALT or AST elevated more than 2 times the upper limits;
3. not well controlled diabetes;
4. uncontrolled heart failure od renal dysfunction(eGFR<30ml/min);
5. Patients with active infection,including tuberculosis, hepatitis B and C,HIV infection, bacteria or fungal infection;
6. upper GI bleeding 3 months before enrolement;
7. refractory hypertension;
8. Pregnant or intended to be pregnant 3 months after the trial;
9. Severe coronary artery involvement demonstrated by CTA;
10. severe cranial or cervical or renal artery diseases that need surgery;
11. Patients that should not be included by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-01-05 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
percentage of patients with complete response | week 78
  percentage of patients with complete response at week 78

SECONDARY OUTCOMES:
percentage of patients with partial response | week 78
  percentage of patients with partial response at week 78
Percentage of patients with image progression at the end of study | week 78
  percentage of patients with progress disease demonstrated by CTA or Doppler at week 78
adverse events | 78 weeks
  safety profile of both Adalimumab and Tofacitinib treatment group
intervention procedures | 78 weeks
  percentage of patients who require intervention procedures during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofeng Zeng, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (4):
- China (4):
  - Beijing Anzhen Hospital, Beijing
  - The General Hospital of the People's Liberation Army, Beijing
  - Beijing Shijitan Hospital, Beijing
  - Beijing Xuanwu Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No